CLINICAL TRIAL: NCT05490836
Title: Peginterferon Alfa-2b Combined With Tenofovir Alafenamide Improves the Functional Cure Rate in Patients With HBeAg Negative Chronic Hepatitis B: an Open-labeled, Multicenter, Randomized and Controlled Clinical Study
Brief Title: Functional Cure Rate of Peg-IFNα-2b Combined With TAF in HBeAg Negative CHB Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jiming Zhang, Chief physician, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2022-517
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Chronic Hepatitis B
Keywords: Peg-IFN; Chronic hepatitis B; Functional cure rate
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- continuous treatment arm (Active Comparator)
  Interventions: Biological: PEG IFN α-2b; TAF
- pulse treatment arm (Experimental)
  Interventions: Biological: PEG IFN α-2b; TAF

INTERVENTIONS:
Biological: PEG IFN α-2b; TAF — TAF was orally administered once a day, and PEG IFN α-2b was subcutaneously injected 135 μg or 180μg once a week. treatment continuous for 48 weeks.
  Arms: continuous treatment arm
Biological: PEG IFN α-2b; TAF — TAF was orally administered once a day, and PEG IFN α-2b was subcutaneously injected 135 μg or 180μg once a week for 8 weeks and followed by 4 weeks off. treatment continuous for 48 weeks.
  Arms: pulse treatment arm

SUMMARY:
The study is aimed to explore the safety and efficacy of the pulse usage , comparing to continuous usage, of Peginterferon alfa-2b Injection (PEG IFN α-2b) Combined With tenofovir alafenamide (TAF) in treatment of naive chronic hepatitis B patients with HBeAg negative.

DETAILED DESCRIPTION:
Using antiviral drugs with different mechanisms of action is one of the effective means to improve the therapeutic outcome at present. At the same time, PEG-IFN is currently recognized as the only drug that can improve the functional cure rate of chronic hepatitis B, and PEG-IFN clinical application is limited due to adverse reactions. Exploring ways to reduce adverse reactions of PEG-IFN and improve PEG-IFN curative effects is the hot spot topic but also difficult at present.

Previously clinical practice have found that the temporary withdrawal of interferon have little influences on the whole clinical outcome in patients withdrawal of interferon due to adverse reactions, and there is indeed a continuous effect after the withdrawal of PEG-IFN for a certain period of time. Therefore, it is conceive that pulse usage of PEG-IFN (eg. use for 8 weeks followed by 4 weeks off) may be a effective method to reduce PEG-IFN adverse reactions while ensuring efficacy.

By comparing the safety and efficacy of pulsed and continuous combination therapy of Peg-IFNα-2b with TAF and in treatment naive HBeAg-negative CHB patients, the investigators hope to develop a better treatment plan for chronic hepatitis B.

ELIGIBILITY:
Inclusion criteria:

* Aged between 18 and 65,included.
* HBsAg positive, HBeAg negative, anti HBE antibody positive, HBV-DNA ≥ 2x10^3 IU/ml, ALT is continuously or repeatedly abnormal, or there is definite inflammation, necrosis and / or fibrosis (≥ G2/S2) confirmed in liver biopsy.
* Received no antiviral treatment previously.
* pregnancy test of Female subjects of childbearing must be negative before the enrollment, and all potential subjects must agree to take effective contraceptive measures during the treatment period and within half a year after the end of the treatment.
* Understand and sign the informed consent voluntarily.

Exclusion criteria:

* Known allergy to interferon, nucleos(t)ide drugs, or any ingredient of the drug.
* Currently co-infection with HAV, HCV, HDV, HEV, HIV, or any other virus.
* Cirrhosis or Child-Pugh score of 7 or above.
* Liver disease caused by other reasons (eg. autoimmune liver disease, alcoholic liver disease, nonalcoholic fatty liver disease, drug-induced hepatitis, hepatolenticular degeneration, etc.).
* Pregnant or lactating women.
* Alcoholism or drug abuse within one year prior to the screening.
* Neutrophil count<1.5×10^9/L, hemoglobin<100g/L, or platelet count<80×10^9/L.
* Serum creatinine was higher than the upper limit of normal at screening.
* History of serious disease in heart, brain, kidney, retina, muscle, or other major organ and systems.
* Have a history of mental illness or family history of mental illness, or Hamilton Depression Scale score ≥ 7 points.
* Have a history of endocrine system or autoimmune diseases, such as thyroid disease, systemic lupus erythematosus, sarcoidosis, autoimmune thrombocytopenic purpura, psoriasis, etc.
* Chronic diseases requiring long-term treatment, such as uncontrolled hypertension, diabetes, chronic obstructive pulmonary disease, etc.
* Malignant tumor.
* Suspected hepatocellular carcinoma in B-ultrasound at screening; or fetoprotein alpha was greater than 100ng/ml, or cannot remain stable within 3 months before screening.
* Accepted organ transplantation previously.
* Other reasons that the investigator considers unsuitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The rate of HBsAg negative | week 48

SECONDARY OUTCOMES:
change in HBsAg level from baseline | week 48
The Rate of HBsAg seroconversion | week 48
Proportion of patients with HBV DNA Below the detection limit | week 24 and week 48
Number of patients with treatment-related adverse events | from baseline to week 48